CLINICAL TRIAL: NCT04155853
Title: Distraction Versus Interposition Arthroplasty for Thumb Carpometacarpal Joint Osteoarthritis: A Randomized Controlled Trial
Brief Title: Distraction vs Interposition Arthroplasty for Basilar Thumb Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Dimitrios Kitridis, Principal Investigator, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 597/2019
Record Dates: First submitted 2019-11-04; First posted 2019-11-07 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Thumb Osteoarthritis
Keywords: trapeziectomy; fascia lata; interposition

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interposition Arthroplasty (Active Comparator): Fascia lata interposition arthroplasty for the treatment of thumb carpometacarpal joint osteoarthritis
  Interventions: Procedure: Interposition Arthroplasty
- Hematoma and Distraction Arthroplasty (Active Comparator): Hematoma and Distraction Arthroplasty for the treatment of thumb carpometacarpal joint osteoarthritis
  Interventions: Procedure: Hematoma and Distraction Arthroplasty

INTERVENTIONS:
Procedure: Interposition Arthroplasty — A typical Wagner incision will be used at the thenar skin one centimeter distal to the radial styloid. The interval between the abductor pollicis longus and the extensor pollicis brevis will be developed, while protecting the dorsal sensory branches of the radial nerve. A longitudinal capsulotomy will be performed and after identifying the carpometacarpal and scaphotrapeziotrapezoid joints, the trapezium will be excised. Then, the empty space will be filled with a roll of fascia lata and fixed with a K-wire. The 1.4 millimeter K-wire will be introduced two centimeters distally to the metacarpal base and into the body of the trapezium. In case of scaphotrapeziotrapezoid joint arthritis, debridement and osteophyte excision of the scaphotrapezoid joint will be performed. In the end of the procedure, the capsule and the skin will be sutured, and a thumb spica will be placed to all patients.
  Arms: Interposition Arthroplasty
Procedure: Hematoma and Distraction Arthroplasty — A typical Wagner incision will be used at the thenar skin one centimeter distal to the radial styloid. The interval between the abductor pollicis longus and the extensor pollicis brevis will be developed, while protecting the dorsal sensory branches of the radial nerve. A longitudinal capsulotomy will be performed and after identifying the carpometacarpal and scaphotrapeziotrapezoid joints, the trapezium will be excised. Then, the empty space will be stabilized with a K-wire without interposition of any material. The 1.4 millimeter K-wire will be introduced two centimeters distally to the metacarpal base and into the body of the trapezium. In case of scaphotrapeziotrapezoid joint arthritis, debridement and osteophyte excision of the scaphotrapezoid joint will be performed. In the end of the procedure, the capsule and the skin will be sutured, and a thumb spica will be placed to all patients.
  Arms: Hematoma and Distraction Arthroplasty

SUMMARY:
Surgical management for osteoarthritis of the thumb is indicated when conservative measures have failed, and numerous techniques have been proposed. Distraction arthroplasty has been the gold standard due to lack of high quality evidence, which renders the benefits or harms of other techniques uncertain. The other treatment alternatives share at least partial excision of the trapezium, and include ligament reconstruction alone or with tendon interposition, allograft interposition arthroplasty, prosthetic implants and arthrodesis. A recent promising technique is the pillow technique, a type of interposition arthroplasty, which utilizes a fascia lata allograft as interposition material and stabilization with a K-wire.

In view of the low quality evidence regarding the use of interposition material versus distraction arthroplasty alone, the investigators will compare the two methods in a prospective randomized study design. Hypothesis of the study is that interposition arthroplasty using the pillow technique yields better results in terms of functional improvement and grip strength when compared to the hematoma and distraction technique. The confirmation of the hypothesis is going to justify the use of the fascia lata in the procedure. On the contrary, if the pillow technique fails to yield clinically meaningful results, the recommendation of the hematoma and distraction technique will account for reducing the overall cost of the procedure, rendering the allograft redundant.

DETAILED DESCRIPTION:
Osteoarthritis is a degenerative disease of the joints, mostly known for the hip and the knee. Osteoarthritis of the thumb carpometacarpal joint is a common cause for pain, stiffness and grip weakness of the hand, affecting one of three females and one of eight males. Surgical management is indicated when conservative measures have failed, and numerous techniques have been proposed. Distraction arthroplasty has been the gold standard due to lack of high quality evidence, which renders the benefits or harms of other techniques uncertain. A recent Cochrane review was unable to demonstrate whether any technique confers a benefit over distraction arthroplasty and noted that the quality of evidence was low.

Hematoma arthroplasty includes trapeziectomy without interposition of any material or ligament reconstruction. Later, the same technique with the addition of a temporary K-wire stabilization of the first metacarpal has been described it as hematoma and distraction arthroplasty. They immobilized the metacarpal in an overcorrected position to avoid postoperative weakness, assuming the causative factor was the subsidence of the metacarpal into the trapezial void, and they reported improved outcomes. The other treatment alternatives share at least partial excision of the trapezium, and include ligament reconstruction alone or with tendon interposition, allograft interposition arthroplasty, prosthetic implants and arthrodesis. A recent promising technique is the pillow technique, a type of interposition arthroplasty, which utilizes a fascia lata allograft as interposition material and stabilization with a K-wire. The technique showed promising results in a long-term follow-up study, and proved to be a viable alternative to distraction arthroplasty with no donor site morbidity and better preservation of the height of the metacarpal. However, there is no robust evidence that retaining the joint space affects the functional results or the grip strength of the patients.

Aim of the study In view of the low quality evidence regarding the use of interposition material versus distraction arthroplasty alone, the investigators will compare the two methods in a prospective randomized study design. Hypothesis of the study is that interposition arthroplasty using the pillow technique yields better results in terms of functional improvement and grip strength when compared to the hematoma and distraction technique. The confirmation of the hypothesis is going to justify the use of the fascia lata in the procedure, which is one option widely utilized. On the contrary, if the pillow technique fails to yield clinically meaningful results, the recommendation of the hematoma and distraction technique will account for reducing the overall cost of the procedure, rendering the allograft redundant.

The study will be conducted in accordance with the Declaration of Helsinki and the Guidelines on Good Clinical Practice.

ELIGIBILITY:
Inclusion Criteria:

* Thumb carpometacarpal osteoarthritis Stage III and IV according to the Eaton and Littler classification
* At least one month history of pain refractory to nonoperative treatment (rest, non-steroidal anti-inflammatory medicine, splint, hand therapy, a maximum of three corticosteroid injections)
* Patient willing to participate to the study

Exclusion Criteria:

* Previous operation to the affected area
* Pregnant patient
* Chronic systemic illnesses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2019-04-16 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
"Quick Disabilities of the Arm, Shoulder, and Hand" (QuickDASH) functional score | six months
  Comparison of the Quick DASH score between the groups. Minimum 0, Maximum 100, higher scores mean a worse outcome.
"Quick Disabilities of the Arm, Shoulder, and Hand" (QuickDASH) functional score | one year
  Comparison of the Quick DASH score between the groups. Minimum 0, Maximum 100, higher scores mean a worse outcome.
"Quick Disabilities of the Arm, Shoulder, and Hand" (QuickDASH) functional score | two years
  Comparison of the Quick DASH score between the groups. Minimum 0, Maximum 100, higher scores mean a worse outcome.
"Visual Analog Scale" (VAS) for pain relief | six months
  Comparison of the VAS for pain between the groups. Minimum 0, Maximum 100, higher scores mean a worse outcome.
"Visual Analog Scale" (VAS) for pain relief | one year
  Comparison of the VAS for pain between the groups. Minimum 0, Maximum 100, higher scores mean a worse outcome.
"Visual Analog Scale" (VAS) for pain relief | two years
  Comparison of the VAS for pain between the groups. Minimum 0, Maximum 100, higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Thumb range of motion (ROM) | six months
  Comparison of thumb ROM between the groups. Flexion, extension, and abduction will be measured for thumb carpometacarpal and interphalangeal joints using a goniometer.
Thumb range of motion (ROM) | one year
  Comparison of thumb ROM between the groups. Flexion, extension, and abduction will be measured for thumb carpometacarpal and interphalangeal joints using a goniometer.
Thumb range of motion (ROM) | two years
  Comparison of thumb ROM between the groups. Flexion, extension, and abduction will be measured for thumb carpometacarpal and interphalangeal joints using a goniometer.
Kapandji score for thumb opposition | six months
  Comparison of the Kapandji score between the groups. Minimum 0, Maximum 10, higher scores mean a better outcome
Kapandji score for thumb opposition | one year
  Comparison of the Kapandji score between the groups. Minimum 0, Maximum 10, higher scores mean a better outcome
Kapandji score for thumb opposition | two years
  Comparison of the Kapandji score between the groups. Minimum 0, Maximum 10, higher scores mean a better outcome

OTHER OUTCOMES:
Rate of complications | Up to two years postoperatively
  All complications will be documented and rates will be compared between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis Givissis, Professor, Study Director — Aristotle University Of Thessaloniki
Locations (1):
- "George Papanikolaou" Hospital, Thessaloniki, Exohi, Greece

REFERENCES:
- [Background] Sodha S, Ring D, Zurakowski D, Jupiter JB. Prevalence of osteoarthrosis of the trapeziometacarpal joint. J Bone Joint Surg Am. 2005 Dec;87(12):2614-2618. doi: 10.2106/JBJS.E.00104. PMID 16322609
- [Background] Martou G, Veltri K, Thoma A. Surgical treatment of osteoarthritis of the carpometacarpal joint of the thumb: a systematic review. Plast Reconstr Surg. 2004 Aug;114(2):421-32. doi: 10.1097/01.prs.0000131989.86319.b1. PMID 15277809
- [Background] Wajon A, Vinycomb T, Carr E, Edmunds I, Ada L. Surgery for thumb (trapeziometacarpal joint) osteoarthritis. Cochrane Database Syst Rev. 2015 Feb 23;2015(2):CD004631. doi: 10.1002/14651858.CD004631.pub4. PMID 25702783
- [Background] Gervis WH, Wells T. A review of excision of the trapezium for osteoarthritis of the trapezio-metacarpal joint after twenty-five years. J Bone Joint Surg Br. 1973 Feb;55(1):56-7. No abstract available. PMID 4693892
- [Background] Kuhns CA, Emerson ET, Meals RA. Hematoma and distraction arthroplasty for thumb basal joint osteoarthritis: a prospective, single-surgeon study including outcomes measures. J Hand Surg Am. 2003 May;28(3):381-9. doi: 10.1053/jhsu.2003.50078. PMID 12772092
- [Background] Givissis P, Sachinis NP, Akritopoulos P, Stavridis SI, Christodoulou A. The "Pillow" Technique for Thumb Carpometacarpal Joint Arthritis: Cohort Study With 10- to 15-Year Follow-Up. J Hand Surg Am. 2016 Jul;41(7):775-81. doi: 10.1016/j.jhsa.2016.04.018. Epub 2016 May 21. PMID 27215594
- [Background] Heller GZ, Manuguerra M, Chow R. How to analyze the Visual Analogue Scale: Myths, truths and clinical relevance. Scand J Pain. 2016 Oct;13:67-75. doi: 10.1016/j.sjpain.2016.06.012. Epub 2016 Jul 27. PMID 28850536
- [Background] Dworkin RH, Turk DC, Farrar JT, Haythornthwaite JA, Jensen MP, Katz NP, Kerns RD, Stucki G, Allen RR, Bellamy N, Carr DB, Chandler J, Cowan P, Dionne R, Galer BS, Hertz S, Jadad AR, Kramer LD, Manning DC, Martin S, McCormick CG, McDermott MP, McGrath P, Quessy S, Rappaport BA, Robbins W, Robinson JP, Rothman M, Royal MA, Simon L, Stauffer JW, Stein W, Tollett J, Wernicke J, Witter J; IMMPACT. Core outcome measures for chronic pain clinical trials: IMMPACT recommendations. Pain. 2005 Jan;113(1-2):9-19. doi: 10.1016/j.pain.2004.09.012. No abstract available. PMID 15621359
- [Background] Smith MV, Calfee RP, Baumgarten KM, Brophy RH, Wright RW. Upper extremity-specific measures of disability and outcomes in orthopaedic surgery. J Bone Joint Surg Am. 2012 Feb 1;94(3):277-85. doi: 10.2106/JBJS.J.01744. PMID 22298061
- [Background] Calfee RP, Adams AA. Clinical research and patient-rated outcome measures in hand surgery. J Hand Surg Am. 2012 Apr;37(4):851-5. doi: 10.1016/j.jhsa.2012.01.043. PMID 22464236
- [Background] Kapandji A. [Clinical test of apposition and counter-apposition of the thumb]. Ann Chir Main. 1986;5(1):67-73. doi: 10.1016/s0753-9053(86)80053-9. French. PMID 3963909
- [Background] Eaton RG, Littler JW. Ligament reconstruction for the painful thumb carpometacarpal joint. J Bone Joint Surg Am. 1973 Dec;55(8):1655-66. No abstract available. PMID 4804988
- [Background] Vermeulen GM, Brink SM, Slijper H, Feitz R, Moojen TM, Hovius SE, Selles RW. Trapeziometacarpal arthrodesis or trapeziectomy with ligament reconstruction in primary trapeziometacarpal osteoarthritis: a randomized controlled trial. J Bone Joint Surg Am. 2014 May 7;96(9):726-33. doi: 10.2106/JBJS.L.01344. PMID 24806009
- [Background] Barthel L, Hidalgo Diaz JJ, Vernet P, Gouzou S, Facca S, Igeta Y, Liverneaux P. Results of the treatment of first carpometacarpal joint osteoarthritis: trapeziectomy alone versus trapeziectomy associated with suspensionplasty. Eur J Orthop Surg Traumatol. 2018 Dec;28(8):1555-1561. doi: 10.1007/s00590-018-2173-3. Epub 2018 Mar 7. PMID 29516197
- [Background] Dupont WD, Plummer WD Jr. Power and sample size calculations. A review and computer program. Control Clin Trials. 1990 Apr;11(2):116-28. doi: 10.1016/0197-2456(90)90005-m. PMID 2161310
- [Background] Nicholson RH, Crawley FP. Revising the Declaration of Helsinki: a fresh start. Bull Med Ethics. 1999 Oct;No. 151:13-7. No abstract available. PMID 11657985